CLINICAL TRIAL: NCT00904293
Title: Randomized Controlled Trial of Genotype-Guided Dosing of Warfarin Therapy
Brief Title: Genotype-Guided Warfarin Therapy Trial
Acronym: WARFPGX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: UNC Institute for Pharmacogenomics and Individualized Therapy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-1644
Record Dates: First submitted 2009-04-06; First posted 2009-05-19 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2013-10

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Pulmonary Embolism; Artificial Heart Valve
Keywords: warfarin; CYP2C9; VKOR; Coumadin; pharmacogenetics; pharmacogenomics; anticoagulation; genotype-guided therapy
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Genotype-guided warfarin dosing (Experimental): A dosing algorithm including clinical factors and genotype information (VKORC1 and CYP2C9) will be used to determine initial warfarin doses.
  Interventions: Other: Genotype-guided dose determination
- Non-genotype guided warfarin dosing (Active Comparator): Initial warfarin dosing will be determined using the same algorithm as in the experimental group, but only including the clinical factors and not including the genotype information
  Interventions: Other: Non-genotype guided warfarin dosing

INTERVENTIONS:
Other: Genotype-guided dose determination — Patients in both arms will be treated with warfarin. Those in the experimental group will have initial doses determined using an algorithm (from www.warfarindosing.org) incorporating genetic and clinical factors. Those in the control group will have doses determined using the same algorithm, but without including the genetic factors.
  Arms: Genotype-guided warfarin dosing
Other: Non-genotype guided warfarin dosing — Those in the control group will have doses determined using the same algorithm, but without including the genetic factors.
  Arms: Non-genotype guided warfarin dosing

SUMMARY:
The purpose of the investigators' study is to determine the clinical utility of a warfarin-dosing algorithm that incorporates genetic information (VKORC1 and CYP2C9 alleles) for adult patients initiating warfarin therapy.

DETAILED DESCRIPTION:
Almost 20 million prescriptions are written for warfarin each year in the US and yet it is one of the most problematic drugs in the modern medical formulary. Warfarin has a narrow therapeutic window and the hemorrhagic or thrombotic implications of modest over- or under-dosing can be devastating. Warfarin is one of the leading causes of emergency department visits and hospitalizations due to adverse drug events worldwide. Adverse events from warfarin are more common during the initial months of treatment before the optimal dose is determined. Moreover, there is substantial individual variation in response to warfarin necessitating frequent monitoring and dosage adjustments. The monitoring and dosing of warfarin is so problematic that many primary care physicians have abdicated this role to specialized "warfarin clinics" which are devoted solely to following patients on this agent. Unfortunately, no good alternatives to warfarin exist for the common indications requiring chronic anticoagulation such as atrial fibrillation, deep vein thrombosis, pulmonary embolism, and artificial heart valves.

Pharmacogenomics offers substantial hope for improved care of patients taking warfarin. One group estimated that formally integrating genetic testing into routine warfarin therapy in the US could result in the avoidance of 85,000 serious bleeding events and 17,000 strokes annually with a cost savings of over $1 billion annually. Common single nucleotide polymorphisms (SNPs) in the gene encoding Vitamin K Epoxide Reductase (VKOR) substantially affect one's sensitivity to warfarin, mediating a doubling or halving of the dose required for optimal anticoagulation. Warfarin inhibits clotting by inhibiting the enzyme VKOR, and thus inhibiting vitamin K dependent clotting factors. A number of recent retrospective studies have shown that polymorphisms in the VKOR gene may account for 20-30% of the variance in warfarin dose seen in patients on stable, long-term warfarin therapy.

Another genetic determinant of variance in warfarin dose is the cytochrome p450 2C9 enzyme CYP2C9. It is almost wholly responsible for metabolism of the more active S-enantiomer of warfarin. The 2C9*2 and 2C9*3 polymorphisms in the CYP2C9 gene are associated with reduced warfarin metabolism, and a number of retrospective studies have shown that these polymorphisms may account for 10-15% of the variance in warfarin dosage in patients on stable, long-term warfarin therapy. In addition, the variant CYP2C9 alleles have been associated with longer times to stabilization of INR and a higher risk for bleeding events. These polymorphisms are seen in ~20-30% of the Caucasian population, but are rare in African Americans and Asians. Together, known VKOR and CYP2C9 variants may account for 40% of the variability in warfarin dosing.

By combining clinical information such as weight, height, and concomitant medications with VKOR and CYP2C9 genotypic information, several algorithms have been devised that calculate warfarin doses. These algorithms have been shown to accurately predict warfarin doses in retrospective studies of patients already on long-term stable warfarin doses. Some small, pilot studies in orthopedic patients suggest that prospective genetic-based dosing is feasible and may result in achieving stable doses sooner in patients with certain genetic variants. However, the prospective studies are small, pilot studies limited to orthopedic patients that did not include medical patients with common indications requiring chronic oral anticoagulation. They are also limited by study designs that include only historical controls. No RCTs have been reported in the literature and further evaluation is needed to determine the utility and cost-effectiveness of genetic-based algorithms. The NHLBI is planning a double-blind, randomized three-arm trial, but the trial will not begin enrolling subjects until 2008 at the earliest and data analysis and dissemination is planned to begin beyond 2011.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* Patients who are beginning warfarin for a variety of diseases or conditions that require long-term oral anticoagulation with target INR > 2.0 for at least 3 months
* Subjects that will be following up in UNC anticoagulation clinics at the Ambulatory Care Center or the Family Medicine Center

Exclusion Criteria:

* Patients who are unable to complete the study materials (questionnaires) with or without assistance (for example, those with dementia)
* Non-English speaking patients
* Patients who are being started on anticoagulation intended to last < 3 months or whose target INR is < 2.0
* Patients who have a history of treatment with warfarin and a known dose requirement will be excluded (as they should be restarted on the previous dose)
* Pregnant women will be excluded because warfarin is a teratogen and pregnant women should not take the medication
* Patients will also be excluded if their treating physician does not agree to use the recommended INR dose or feels that the patient should not be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Time in therapeutic range (TTR) | 3 months
Number of anticoagulation visits | 3 months

SECONDARY OUTCOMES:
Proportion of INRs > 4 | 3 months
Major bleeding events | 3 months
Minor bleeding events | 3 months
Thromboembolic complications | 3 months
All-cause mortality | 3 months
Time to therapeutic dose | 3 months
Emergency department visits | 3 months
Hospitalizations | 3 months
Costs and cost-effectiveness | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Jonas, MD, MPH, Principal Investigator — UNC Institute for Pharmacogenomics and Individualized Therapy
Locations (1):
- UNC Hospitals, UNC Anticoagulation Clinic at the Ambulatory Care Center (ACC), UNC Family Medicine Center Anti-coagulation Clinic, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Levine MN, Raskob G, Landefeld S, Kearon C. Hemorrhagic complications of anticoagulant treatment. Chest. 2001 Jan;119(1 Suppl):108S-121S. doi: 10.1378/chest.119.1_suppl.108s. PMID 11157645
- [Background] Hafner JW Jr, Belknap SM, Squillante MD, Bucheit KA. Adverse drug events in emergency department patients. Ann Emerg Med. 2002 Mar;39(3):258-67. doi: 10.1067/mem.2002.121401. PMID 11867978
- [Background] McWilliam A, Lutter R, Nardinelli C. Jointcenter; AEI-Brookings Joint Center For Regulatory Studies. Working Paper 06-23, November 2006
- [Background] Rieder MJ, Reiner AP, Gage BF, Nickerson DA, Eby CS, McLeod HL, Blough DK, Thummel KE, Veenstra DL, Rettie AE. Effect of VKORC1 haplotypes on transcriptional regulation and warfarin dose. N Engl J Med. 2005 Jun 2;352(22):2285-93. doi: 10.1056/NEJMoa044503. PMID 15930419
- [Background] Li T, Lange LA, Li X, Susswein L, Bryant B, Malone R, Lange EM, Huang TY, Stafford DW, Evans JP. Polymorphisms in the VKORC1 gene are strongly associated with warfarin dosage requirements in patients receiving anticoagulation. J Med Genet. 2006 Sep;43(9):740-4. doi: 10.1136/jmg.2005.040410. Epub 2006 Apr 12. PMID 16611750
- [Background] Sconce EA, Khan TI, Wynne HA, Avery P, Monkhouse L, King BP, Wood P, Kesteven P, Daly AK, Kamali F. The impact of CYP2C9 and VKORC1 genetic polymorphism and patient characteristics upon warfarin dose requirements: proposal for a new dosing regimen. Blood. 2005 Oct 1;106(7):2329-33. doi: 10.1182/blood-2005-03-1108. Epub 2005 Jun 9. PMID 15947090
- [Background] Millican, E., et al. Blood, Epub ahead of print, Mar 26, 2007
- [Background] Voora D, Eby C, Linder MW, Milligan PE, Bukaveckas BL, McLeod HL, Maloney W, Clohisy J, Burnett RS, Grosso L, Gatchel SK, Gage BF. Prospective dosing of warfarin based on cytochrome P-450 2C9 genotype. Thromb Haemost. 2005 Apr;93(4):700-5. doi: 10.1160/TH04-08-0542. PMID 15841315
- [Derived] Jonas DE, Evans JP, McLeod HL, Brode S, Lange LA, Young ML, Shilliday BB, Bardsley MM, Swinton-Jenkins NJ, Weck KE. Impact of genotype-guided dosing on anticoagulation visits for adults starting warfarin: a randomized controlled trial. Pharmacogenomics. 2013 Oct;14(13):1593-603. doi: 10.2217/pgs.13.145. PMID 24088130